CLINICAL TRIAL: NCT01860274
Title: External Mesh of Vein Grafts In Coronary Artery Bypass Grating: Early Patency and Clinical Outcome
Brief Title: Meshed Vein Graft Patency Trial - VEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-06
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
Keywords: Mesh; Graft; Patency
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- External Mesh (Experimental)
  Interventions: Device: External Mesh for vein grafts

INTERVENTIONS:
Device: External Mesh for vein grafts

SUMMARY:
The study hypothesis is that a meshed conduit made of safen vein allows a better patency at mid-long term than a safen vein alone.

To test this hypothesis the investigators plan a prospective, randomized study, comparing grafts to the diagonal, in cases of vessel diameter under 1.5mm. A control angiography will be performed one year after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Indication for elective Coronary Artery Bypass Grafting with at least one vein graft
* Coronary artery with critical stenosis (over 70%)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-09-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Patency | 6 to 12 months
  Patency of graft at CT Scan

SECONDARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 60 months
Vein graft lumen uniformity | 6 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Luca Weltert, MD, Principal Investigator — European Hospital - Rome; Ruggero De Paulis, MD, Study Chair — European Hospital - Rome
Locations (2):
- Italy (2):
  - European Hospital, Rome
  - Mauriziano Hospital, Turin

REFERENCES:
- [Derived] Weltert LP, Audisio K, Bellisaro A, Bardi G, Flocco R, De Paulis R, Centofanti P. External stenting of vein grafts in coronary artery bypass grating: interim results from a two centers prospective study. J Cardiothorac Surg. 2021 Apr 12;16(1):74. doi: 10.1186/s13019-021-01406-0. PMID 33845865